CLINICAL TRIAL: NCT03576105
Title: Evaluation of Photodynamic Therapy in Pericoronitis: a Randomized, Controlled, Double-blind Clinical Study
Brief Title: Evaluation of Photodynamic Therapy in Pericoronitis
Acronym: pdt
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Anna Carolina Ratto Tempestini Horliana, Clinical Professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: pericoronitis
Record Dates: First submitted 2018-06-06; First posted 2018-07-03 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Pericoronitis
Keywords: third molar; pericoronitis; photodynamic therapy; microbiological analysis; laser; randomized controlled clinical study
MeSH Terms: conditions — Pericoronitis | interventions — Therapeutic Irrigation; Photosensitizing Agents; Photochemotherapy; Methylene Blue; 1-phenyl-3,3-dimethyltriazene

STUDY DESIGN:
Intervention Model Description: Endpoint Classification: Bio-equivalence Study Enrollment: 34 [Anticipated]
Who Masked: Participant, Investigator
Masking Description: Double Blind (Subject, Caregiver, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): G1 - 17 patients Photodynamic therapy with convention methylene blue as photosesintizer irrigation /sterile saline Conventional methylene blue as photosensitizer -Irrigation with 0,04mL of photosensitizer (0,005%) inside the gingival sulcus around the third molar with pericoronarite for 3 minutes Photodynamic therapy -Device irradiation with low intensity laser λ = 660 nm, 9J per point and radiant 90 seconds
  Interventions: Combination Product: irrigation /sterile saline; Combination Product: Conventional methylene blue as photosensitizer; Combination Product: Photodynamic therapy
- positive control group (Active Comparator): G2 - 17 patients Photodynamic therapy with oral formula of methylene blue as photosesintizer, treatment identical to G1, however methylene blue will be delivered in a new formulation for oral use (patent aplicattion INPI BR1020170253902) irrigation /sterile saline Photodynamic therapy -Methylene blue for oral use as photosensitizer-Irrigation with 0,04mL of photosensitizer (0,005%) inside the gingival sulcus around the third molar with pericoronarite for 3 minutes Device irradiation with low intensity laser λ = 660 nm, 9J per point and radiant 90 seconds
  Interventions: Combination Product: irrigation /sterile saline; Combination Product: Methylene blue for oral use as photosensitizer; Combination Product: Photodynamic therapy

INTERVENTIONS:
Combination Product: irrigation /sterile saline — mechanical removal of bacteria with sterile saline
Combination Product: Conventional methylene blue as photosensitizer — Irrigation with 0,04mL of photosensitizer (0,005%) inside the gingival sulcus around the third molar with pericoronarite for 3 minutes
  Other Names: photodynamic therapy with conventional methylene blue
  Arms: experimental group
Combination Product: Methylene blue for oral use as photosensitizer — Irrigation with 0,04mL of photosensitizer(0,005%) inside the gingival sulcus around the third molar with pericoronarite for 3 minutes
  Other Names: photodynamic therapy with methylene blue for oral use
  Arms: positive control group
Combination Product: Photodynamic therapy — Red laser for photodynamic therapy (Therapy XT,DMC,Sao Carlos,Sao Paulo,Brazil) Device irradiation with low intensity laser λ = 660 nm, 9J per point and radiant 90 seconds
  Other Names: PDT

SUMMARY:
In order to reduce the chances of systemic dissemination of the infection and the use of antibiotics, it is mandatory to test effective treatments in the initial phase of pericoronitis aiming to avoid the evolution of the infectious disease. Photodynamic therapy (PDT) is an interesting alternative because it is an effective antimicrobial treatment that is easy to perform and does not cause bacterial resistance. The aim of this study is to evaluate the effectiveness of photodynamic therapy (PDT) with methylene blue in a surfactant vehicle in pericoronitis in the initial phase in healthy youngsters through microbiological, clinical and immunoregulatory response. The impact of pericoronitis on oral health-related quality of life (OHRQoL) of these patients will also be evaluated. 34 healthy young patients with pericoronitis will be evaluated. Microbiological analysis will be performed by RT-PCR for the bacterium Tannarella forsithia (Tf).Gingival crevicular fluid will be collected to evaluate TNF-α, IL1-β, IL-6 and IL-8 and IL-10 by the Luminex assay. The variables will be pain (visual analogue scale), edema, trismus (digital caliper) and oral health-related quality of life (OHRQoL) will also be evaluated through the OHIP-14 questionnaire. The variables will be assessed at T1 (baseline)and T2 (4th day after PDT).

DETAILED DESCRIPTION:
Pericoronitis is a common disease in the eruption phase of third molars, sometimes debilitating, with an impact on the quality of life. The most indicated treatment in the initial phase is the irrigation for cleanliness of the region. If there is no adequate treatment at this stage, there may be evolution of the infectious condition so that antibiotic therapy is indicated. In order to reduce the chances of systemic dissemination of the infection and the use of antibiotics, it is mandatory to test effective treatments in the initial phase of pericoronitis aiming to avoid the evolution of the infectious disease. Photodynamic therapy (PDT) is an interesting alternative because it is an effective antimicrobial treatment that is easy to perform and does not cause bacterial resistance. The methylene blue used in PDT has been studied in a surfactant vehicle, which optimizes the formation of monomers increasing its antimicrobial action. Objective: The aim of this study is to evaluate the effectiveness of photodynamic therapy (PDT) with methylene blue in an surfactant vehicle in pericoronitis in the initial phase in healthy youngsters through microbiological, clinical and immunoregulatory response. The impact of pericoronitis on oral health-related quality of life (OHRQoL) of these patients will also be evaluated. Method: In this randomized, controlled, double-blind clinical bioequivalence trial, 34 healthy young patients with pericoronitis will be evaluated. Patients will be randomized into the positive control group (G1) (n = 17): irrigation with sterile saline and photodynamic therapy (conventional methylene blue at 0.005% concentration and irradiation with low intensity laser λ = 660 nm, 9J per point and radiant exposure of 318 J / cm2), and the experimental group (G2) (n = 17): treatment identical to G1, however methylene blue will be delivered in a new formulation for oral use. Microbiological analysis will be performed by RT-PCR for the bacterium Tannerella forsithia (Tf).Non-stimulated saliva will be collected to evaluate TNF-α, IL1-β, IL-6 and IL-8 and IL-10 by Luminex assay. The pain (visual analogue scale), edema and buccal opening (digital caliper) and oral health-related quality of life (OHRQoL) will also be evaluated through the OHIP-14 questionnaire. The variables will be evaluated in T1 (baseline), and T2 (4th day after PDT).

ELIGIBILITY:
Inclusion Criteria:

* Patients should have at least one lower third partially visible molar in the oral cavity to be examined (Lower third molar erupted or partially erupted, with pericoronitis)
* All patients, regardless of age, gender, cultural level or socioeconomic status may participate in the research.

Exclusion Criteria:

* patients allergic to methylene blue
* pregnant or breastfeeding women,
* those with local infection (e.g., pericoronitis or periodontal abscess) presence of purulent exudate,
* those with fever (temperature above 37.8 C)
* Patients who have used anti-inflammatory drugs or antibiotic medications in the last three months will also be excluded.

Ages: 13 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 34 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2024-04-20 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Microbiological analysis will be performed by RT-PCR for the bacterium Tannarella forsithia (Tf) | change from baseline, immediately after PDT and on fourth day after PDT
  Sample collection for microbiological analysis Biofilm collection will be done at two points of the vestibular gingival sulcus of the lower third molar using minifive curettes. The collected material will be maintained in TE (Tris-EDTA), conditioned in microtubes and later transported for laboratory analysis in the Microbiology Laboratory of ICB-USP Prof. Marcia Mayer

SECONDARY OUTCOMES:
Profile of cytokines Gingival crevicular fluid will be collected | change from baseline and on fourth day after PDT
  gingival crevicular fluid sample will be obtained. Samples will be kept in ice cube tubes. The saliva will be centrifuged at 4000 rpm for 10 minutes at -4 ° C and stored at -80 ° C for further analysis. Determination of plasma levels of the inflammatory markers TNF-α, IL1-β, IL-6 and IL-8 by Luminex assay
pain assessed by Vas | change from baseline, immediately after PDT and on fourth day after PDT
  The pain will be assessed by applying a VAS visual analogic scale, consisting of a 100-mm line numbered in centimeters, with two closed ends. One end is labeled "0" and the other "100", meaning no pain and terrible pain, respectively. Each patient will be instructed to mark a vertical line with the point that best matches the intensity of pain during the evaluation. Instructions on marking will always be given to the patient by the same operator
edema assessed by measuring facial distance | change from baseline, immediately after PDT and on fourth day after PDT
  The criteria for the determination of edema will follow pre-established measurements: (I) Corner of the eye to angle of the jaw (II) Tragus to the labial commissure and (III) Tragus to pogonion as described by Ustun, 2003. Edema will be the sum of three pre-established facial measures (using a digital caliper).
trismus assessed by measuring bucal opening | change from baseline, immediately after PDT and on fourth day after PDT
  For evaluation of the presence of trismus the inter-incisor measurement (distance between the incisal edge of the maxillary central incisor and lower) will be used with a digital caliper (Mitutoyo Digimatic Caliper model, Japan).
OHRQoL assessed by ohip-14 | change from baseline, immediately after PDT and on fourth day after PDT
  Oral health related quality of life: using OHIP-14 questionnaire we will assess the impact on HRQOL will be measured. This instrument consists of 14 items arranged in 7 factors: functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability, and handicap. The answers are given in a 5-point Likert scale (0 = never, 1 = rarely, 2 = sometimes, 3 = often, 4 = always).
position and classification of third molar | baseline
  Position and classification of the lower third molars: the position of the teeth will be assessed by panoramic radiography, according to the classification of Pell and Gregory and Winter (1942), performed only by an evaluator, following the criteria of imaginary lines as proposed by Almendros-Marques , (2008).

CONTACTS AND LOCATIONS:
Overall Officials: Anna Carolina Ratto T Horliana, phd, Principal Investigator — Nove de Julho university (UNINOVE)
Locations (1):
- Nove de Julho University, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] da Silva T, da Silva FC, Gomes AO, Viana AO, Goncalves MLL, Rodrigues MFSD, Horliana ACRT, da Silva DFT, Chavantes MC, Fragoso YD, Branco LP, Motta LJ, Fernandes KPS, Mesquita-Ferrari RA, Bussadori SK. Effect of photobiomodulation treatment in the sublingual, radial artery region, and along the spinal column in individuals with multiple sclerosis: Protocol for a randomized, controlled, double-blind, clinical trial. Medicine (Baltimore). 2018 May;97(19):e0627. doi: 10.1097/MD.0000000000010627. PMID 29742699
- [Background] Sobral APT, Godoy CLH, Fernandes KPS, Bussadori SK, Ferrari RAM, Horliana ACRT, Monken SF, Motta LJ. Photomodulation in the treatment of chronic pain in patients with temporomandibular disorder: protocol for cost-effectiveness analysis. BMJ Open. 2018 May 5;8(5):e018326. doi: 10.1136/bmjopen-2017-018326. PMID 29730613
- [Background] da Cunha Moraes G, Vitoretti LB, de Brito AA, Alves CE, de Oliveira NCR, Dos Santos Dias A, Matos YST, Oliveira-Junior MC, Oliveira LVF, da Palma RK, Candeo LC, Lino-Dos-Santos-Franco A, Horliana ACRT, Gimenes Junior JA, Aimbire F, Vieira RP, Ligeiro-de-Oliveira AP. Low-Level Laser Therapy Reduces Lung Inflammation in an Experimental Model of Chronic Obstructive Pulmonary Disease Involving P2X7 Receptor. Oxid Med Cell Longev. 2018 Mar 4;2018:6798238. doi: 10.1155/2018/6798238. eCollection 2018. PMID 29686745
- [Background] Okamoto CB, Motta LJ, Prates RA, da Mota ACC, Goncalves MLL, Horliana ACRT, Mesquita Ferrari RA, Fernandes KPS, Bussadori SK. Antimicrobial Photodynamic Therapy as a Co-adjuvant in Endodontic Treatment of Deciduous Teeth: Case Series. Photochem Photobiol. 2018 Jul;94(4):760-764. doi: 10.1111/php.12902. Epub 2018 Apr 30. PMID 29420856
- [Background] Belotto RA, Chavantes MC, Tardivo JP, Euzebio Dos Santos R, Fernandes RCM, Horliana ACRT, Pavani C, Teixeira da Silva DF. Therapeutic comparison between treatments for Vulvar Lichen Sclerosus: study protocol of a randomized prospective and controlled trial. BMC Womens Health. 2017 Aug 10;17(1):61. doi: 10.1186/s12905-017-0414-y. PMID 28793884
- [Derived] Schalch TO, Palmieri M, Longo PL, Braz-Silva PH, Tortamano IP, Michel-Crosato E, Mayer MPA, Jorge WA, Bussadori SK, Pavani C, Negreiros RM, Horliana ACRT. Evaluation of photodynamic therapy in pericoronitis: Protocol of randomized, controlled, double-blind study. Medicine (Baltimore). 2019 Apr;98(17):e15312. doi: 10.1097/MD.0000000000015312. PMID 31027098